CLINICAL TRIAL: NCT04386642
Title: Effect of Tranexamic Acid Infusion to Reduce Intraoperative Blood Loss in Large Meningioma: A Prospective Randomized Double-blind Control Study
Brief Title: Tranexamic Acid Reduce Blood Loss in Meningioma Resection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Pathomporn Pin on, M.D., Assistant Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANE_07052020
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Meningioma
Keywords: Tranexamic acid; Meningioma; Blood loss
MeSH Terms: conditions — Meningioma; Hemorrhage | interventions — Tranexamic Acid; Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into two parallel groups by block of four randomization.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and outcome assessors are blinded to the drug that will be prepared by a pharmacist in the similar unlabelled 50-ml syringe.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiment group (Experimental): Each ampule contains TXA 250 mg. TXA preparation is 2000 mg dilute in normal saline 50 ml to get the concentration of 40 mg/ml. TXA will be administered 20 mg/kg loading over 20 min before skin incision followed by a maintenance infusion of 0.025 ml/kg/h (1 mg/kg/h) until the end of operation.
  Interventions: Drug: Tranexamic acid
- Control group (Placebo Comparator): Normal saline solution 50 ml is prepared in a clear 50 ml syringe similar to the experiment group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid 2000 mg dilute in normal saline solution 50 ml.
  Other Names: group T
  Arms: Experiment group
Drug: Placebo — normal saline solution in a clear 50-ml syringe
  Other Names: group N
  Arms: Control group

SUMMARY:
In neurosurgical setting, a large sample size trials of tranexamic acid (TXA) has been limited to TBI and SAH.

The evidence of TXA in brain tumor was scarce. A few case reports support the role of TXA in brain tumor patients with significant intraoperative bleeding and difficult achieving hemostasis. To prove the benefit of TXA for an attenuation of blood loss in brain tumor patients, research with a larger sample size is required. This prospective, randomized double-blind controlled study will be conducted to evaluate the effect of TXA in reducing blood loss and blood transfusion in patients with intracranial meningiomas, diameter > 5 cm in at least 2 dimensions from the latest radiographic findings.

DETAILED DESCRIPTION:
Background and Literature review:

1. Meningioma
2. Coagulation in craniotomy to remove meningioma
3. Bleeding in craniotomy to remove meningioma
4. Tranexamic acid (TXA)
5. Knowledge gap The topics shown above has been reviewed to conduct a prospective randomized double-blind, placebo controlled study.

To prove the study hypothesis: Will intraoperative TXA administration in adult patients scheduled for craniotomy to remove large meningioma decrease blood loss?

ELIGIBILITY:
Inclusion Criteria:

* The patients whose aged 18 to 60 years
* The patients who was diagnosed intracranial meningioma
* The radio-graphic finding of tumor diameter > 5 cm in at least 2 dimensions
* The patients have written informed consent
* The patients is scheduled for elective craniotomy to remove tumor

Exclusion Criteria:

* Patients who refuse to participate in this study
* Patients with recurrent tumor
* The patient is set operation for intracranial tissue biopsy
* The patients with history of TXA allergy
* The pregnant patients
* The patients with history of significant thromboembolic episode
* The patients with significant renal dysfunction (GFR ≤ 50 ml/min)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
volume of intraoperative blood loss | in operating room during surgery
  1. volume of blood presented in the suction bottle subtracted by the amount of water that the surgeon used in the surgical field
  2. the blood from the dry (30 ml) and wet swab (50 ml)
  3. serial Hgb / Hct periodically during surgery and compare to those obtain before surgery

SECONDARY OUTCOMES:
volume of blood being transfused | during surgery and 24 hour after surgery
  volume of pack red cell and other blood component (FFP, platelet)
surgeon rated for the satisfaction on hemostatic scale | in 2 hours after finish the operation
  The surgeon will be informed about a Likert-type scale which is designed for clinical studies. The surgeon's satisfaction on hemostatic scale is a 3-graded scale modified from 5-graded validated bleeding severity scale. The original version is shown in the table 1. The surgeon will judge his satisfaction on hemostatic quality based on the most critical period or the overview of the surgical procedure. Even the long operative time, there will be one rate represent surgeon's opinion on hemostatic quality.
the extent of tumor removal according to the surgeon decision | in 2 hours after finish the operation
  completely or partially resection is rated by the surgeons
postoperative complications | in ICU neuro in 24 hours
  bleeding, remarkable brain edema, re-craniotomy within 24 hours, worsening GCS, DIC, thromboembolic events, postoperative seizures
the duration of postoperative ventilator use | number of day remained intubation within 1 week after surgery
  remain intubation
the length of neuro-ICU stays | number of day remained intubation within 1 week after surgery
  how long the patient stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Pathomporn Pin-on, MD, Principal Investigator — Chiang Mai University
Locations (1):
- Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Ostrom QT, Cioffi G, Gittleman H, Patil N, Waite K, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2012-2016. Neuro Oncol. 2019 Nov 1;21(Supplement_5): v1-v100. doi: 10.1093/neuonc/noz150. 2. Islim, A.I., Mohan, M., Moon, R.D.C. et al. Incidental intracranial meningiomas: a systematic review and meta-analysis of prognostic factors and outcomes. J Neurooncol 142, 211-221 (2019). https://doi.org/10.1007/s11060-019-03104-3 3. Lemée, J., Corniola, M.V., Da Broi, M. et al. Extent of Resection in Meningioma: Predictive Factors and Clinical Implications. Sci Rep 9, 5944 (2019). https://doi.org/10.1038/s41598-019-42451-z 4. Choy W, Kim W, Nagasawa D, Stramotas S, Yew A, Gopen Q, Parsa AT, Yang I. The molecular genetics and tumor pathogenesis of meningiomas and the future directions of meningioma treatments. Neurosurg Focus. 2011 May;30(5): E6. doi: 10.3171/2011.2. FOCUS1116. 5. Sawaya R, Rämö OJ, Shi ML, Mandybur G. Biological significance of tissue plasminogen activator content in brain tumors. J Neurosurg. 1991 Mar;74(3):480-6. 6. Goh KY, Poon WS, Chan DT, Ip CP. Tissue plasminogen activator expression in meningiomas and glioblastomas. Clin Neurol Neurosurg. 2005 Jun;107(4):296-300. 7. Goh KY, Tsoi WC, Feng CS, Wickham N, Poon WS. Haemostatic changes during surgery for primary brain tumours. J Neurol Neurosurg Psychiatry. 1997 Sep;63(3):334-8. 8. J. E. Brecknell, C. A. Mclean, H. Hirano & G. M. Malham. Disseminated intravascular coagulation complicating resection of a malignant meningioma, British Journal of Neurosurgery. 2006, 20:4, 239-241, DOI: 10.1080/02688690600852647 9. Velez AM, Friedman WA. Disseminated intravascular coagulation during resection of a meningioma: case report. Neurosurgery.2011Apr;68(4): E1165-9; discussion E1169.doi: 10.1227/ NEU. 0b013 e31820a18 1a 10. Hsu SY, Huang YH. Characterization and prognostic implications of significant blood loss during intracranial meningioma surgery. Transl Cancer Res 2016;5(6):797-804. doi: 10.21037/tcr.2016.11.72. 11. Wu WC, Trivedi A, Friedmann PD, et al. Association between hospital intraoperative blood transfusion practices for surgical blood loss and hospital surgical mortality rates. Ann Surg 2012; 255:708-14. 12. Tsyben A, Surour M, Budohoski K, et alP42 Predicting bleeding risk during meningioma surgery. Journal of Neurology, Neurosurgery & Psychiatry 2019;90: e35. 13. Yates, J., Perelman, I., Khair, S., Taylor, J., Lampron, J., Tinmouth, A. and Saidenberg, E. (2019), Exclusion criteria and adverse events in perioperative trials of tranexamic acid: a systematic review and meta-analysis. Transfusion, 59: 806-824. doi:10.1111/trf.15030 14. Chauncey JM, Wieters JS. Tranexamic Acid. [Updated 2019 Dec 16]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2020 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK532909/ 15. Shakur H, Roberts I, Bautista R, et al; CRASH-2 trial collaborators. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomized, placebo-controlled trial. Lancet. 2010; 376:23-32. 16. Roberts I, Shakur H, Afolabi A, et al; CRASH-2 collaborators. The importance of early treatment with tranexamic acid in bleeding trauma patients: an exploratory analysis of the CRASH-2 randomized controlled trial. Lancet. 2011; 377:1096- 1101, 1101 e1091-1092. 17. WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomized, double-blind, placebo-controlled trial. Lancet. 2017; 389:2105-2116. 18. Gayet-Ageron A, Prieto-Merino D, Ker K, Shakur H, Ageron FX, Roberts I; Antifibrinolytic Trials Collaboration. Effect of treatment delay on the effectiveness and safety of antifibrinolytics in acute severe haemorrhage: a meta-analysis of individual patient-level data from 40 138 bleeding patients. Lancet. 2018; 391:125-132. 19. Hooda B, Muthuchellappan R. Tranexamic Acid in Neuroanesthesia and Neurocritical Care: Time for Its Critical Appraisal. J Neuroanaesthesiol Crit Care 2019; 6:257-266. 20. Ker K, Prieto-Merino D, Roberts I. Systematic review, meta-analysis and meta-regression of the effect of tranexamic acid on surgical blood loss. Br J Surg 2013;100(10):1271-1279.